CLINICAL TRIAL: NCT06950593
Title: Upper Limb Function Following Transcutaneous Electrical Spinal Cord Stimulation in Individuals With Hemiplegic Stroke
Brief Title: Transcutaneous Electrical Stimulation for Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Mary Ellen Stoykov, Research Scientist, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00220717
Record Dates: First submitted 2025-03-20; First posted 2025-04-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Upper Limb Hemiparesis Following Stroke
Keywords: upper limb hemiparesis; stroke; transcutaneous spinal cord stimulation (TESS)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This interventional study uses a randomized, single-blind (evaluator masked), parallel, two-arm experimental design with an appropriate active comparator.
Who Masked: Participant, Outcomes Assessor
Masking Description: During treatment sessions, both the experimental group and the active comparator group receive the same task specific training protocol as well as don the TESS system. For the active comparator group, the TESS will be turned on to a threshold level of sensation. The participant will be told that the stimulation is being lowered to a below-threshold level, at which point it will be turned off for the rest of the session. This will allow the participants to remain blinded. It is not possible to perform the protocol with blinded treatment therapists. The blinded evaluator is not present during the treatment sessions and will not be told which group the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): This group receives task specific training and transcutaneous spinal cord stimulation (TESS) during treatment sessions. TESS is applied via electrodes placed vertically over the spinous processes of C5-C6. The stimulation will be adjusted within a range of 10mA to 100mA based on participant tolerance and will be delivered for 30 minutes per training session.
  Interventions: Other: Task Specific Training (TST); Other: Transcutaneous electrical spinal cord stimulation (TESS)
- Comparator Group (Active Comparator): This group receives task specific training without real TESS during treatment sessions. Instead, they receive Sham TESS, which is a placebo version in which the electrodes are applied and the stimulation is turned on so that the patient can feel it, and then ramped down to zero for the duration of the session.
  Interventions: Other: Task Specific Training (TST); Other: Sham transcutaneous electrical spinal cord stimulation (Sham TESS)

INTERVENTIONS:
Other: Task Specific Training (TST) — Task specific training activities are types of activities that may be used in standard of care for stroke rehabilitation. Tasks will be completed in sitting or standing. As is usual in studies for upper limb hemiparesis, study participants will be picking up objects with their affected hands. They will work on grasp, grasp-lift of objects, release of objects, reaching and grasping, and reaching without grasping.
Other: Transcutaneous electrical spinal cord stimulation (TESS) — The Digitimer DS8R Transcutaneous Spinal Cord Neurostimulator will deliver transcutaneous electrical spinal cord stimulation. The stimulus intensity used during the intervention will be determined based on individual maximum tolerance. We expect this current amplitude to be between 10mA and 100mA. Stimulation time will be standardized to a 30min duration during which the participant will perform task specific training tasks.
  Arms: Experimental Group
Other: Sham transcutaneous electrical spinal cord stimulation (Sham TESS) — The Sham TESS intervention will utilize the same device and setup as the true TESS intervention. However, after turning on the stimulation and reaching the appropriate intensity, the stimulation will be ramped down and turned off for the remainder of the treatment session. The participant will be told that the stimulation was brought down to a sub-threshold level in order to maintain treatment group blinding.
  Arms: Comparator Group

SUMMARY:
This study aims to evaluate the feasibility and impact of transcutaneous electrical stimulation of the spinal cord (TESS) on the recovery of post-stroke individuals who have upper limb hemiparesis. It will compare outcomes measures between individuals who receive upper limb task specific training with TESS and individuals who receive task specific training of the upper limb with Sham, or fake, TESS.

DETAILED DESCRIPTION:
Upper limb (UL) hemiparesis is the most common post-stroke disability. Currently, there is no treatment used in the clinic that has shown to be efficacious for 75% of individuals who have moderate to severe UL hemiparesis. There are no interventions for individuals with moderate to severe hemiparesis that have demonstrated superiority in comparison to standard care. These stroke patients often have increased spasticity and muscle weakness, resulting in chronic upper limb dysfunction. We are proposing an alternative strategy to improve upper limb function after stroke: transcutaneous electrical stimulation of the spinal cord (TESS). Our objective is to evaluate the feasibility and neural effects of transcutaneous spinal stimulation plus task specific training in a two-arm study with three time points (pre-/post-intervention and follow-up). We will recruit 14 chronic post-stroke participants who will receive 15 sessions of either TESS plus task specific training or Sham TESS plus task specific training. Our long-term research goal is to use TESS as a therapeutic strategy, combined with task specific training, to improve upper limb impairment and function in chronic stroke survivors. Our central hypothesis is that excitation of spinal circuitry by spinal stimulation will result in more effective motor control that will improve volitional upper limb movement (as compared to sham stimulation plus task specific training). This hypothesis is based on published work in cervical spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* able and willing to give written consent and comply with study procedures
* at least 6 months post-stroke
* hemiplegia secondary to stroke
* UE Fugle Meyer Assessment <35
* not currently receiving regular occupational therapy services
* participant has received clearance from physician to participate in study
* participant has at least a rudimentary comprehension of English

Exclusion Criteria:

* botox injection in upper extremity within the last 4 months
* modified ashworth score of 4 in any joint of the affected limb
* pregnant or nursing
* using a powered, implanted cardiac device for monitoring or support of heart function (i.e. pacemaker, defibrillator, or LVAD), or anti-spasticity implantable pumps, or cochlear implants
* unhealed bone fractures
* severe contractures in the upper extremities
* active cancer or cancer remission less than 5 years
* orthopedic dysfunction, injury, or surgery that would impact the individual's ability to use the upper extremities
* recent procedure or operation of the spinal cord within the past year
* traumatic brain injury or neurological conditions that would impact the study
* skull fracture that has developed within the past 6 months
* non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Test of Upper Extremity Function (FMUE) | Session 1 (Week 1): Baseline Evaluation, Session 18 (Week 7): Post-intervention Evaluation, Session 20 (Week 15): Follow-up Evaluation
  The FMUE is an impairment scale that addresses both synergy and isolated movements of the upper limb. The subscales include reflex movements, flexor synergy, extensor synergy, movements out of synergy, combining synergies, wrist, hand, and coordination subscales. The total score ranges from 0 to 66 with higher scores indicating greater function.
Modified Ashworth Scale (MAS) | Session 1 (Week 1): Baseline Evaluation, Session 18 (Week 7): Post-intervention Evaluation, Session 20 (Week 15): Follow-up Evaluation
  The MAS is a test of muscle spasticity and increases in muscle tone. The scores range from 0-4 for each test item, depending on the increase in muscle tone when completing quick movement, or resting muscle tone.
Grip Strength | Session 1 (Week 1): Baseline Evaluation, Session 18 (Week 7): Post-intervention Evaluation, Session 20 (Week 15): Follow-up Evaluation
  Grip strength will be an outcome measure measured via the Jamar Dynamometer. The procedure will consist of 3 tests of maximum grip strength force. Participants will be given ~30 seconds to 1 minute of rest time for each hand in between tests. The individual will maintain ~90 degrees of elbow flexion, 0 degrees of shoulder flexion, and a neutral wrist position while completing the testing.
Chedoke Arm & Hand Activity Index (CAHAI-9) | Session 1 (Week 1): Baseline Evaluation, Session 18 (Week 7): Post-intervention Evaluation, Session 20 (Week 15): Follow-up Evaluation
  The CAHAI 9 is a test of bimanual function. There are nine activities including opening a jar, pouring water, drawing a line with a ruler, buttoning a shirt, using the telephone, wringing out a washcloth, applying toothpaste to a toothbrush, cutting food, and drying one's back with a bath towel. The scale ranges from 1 to 7 for each test item and are graded by the amount of use of the affected hand.
Canadian Occupational Performance Measure (COPM) | Session 1 (Week 1): Baseline Evaluation, Session 18 (Week 7): Post-intervention Evaluation, Session 20 (Week 15): Follow-up Evaluation
  The COPM is a patient-reported outcome measure in which the participant will be asked to rate their ability to perform tasks of everyday living. Specifically, the assessment asks participants to identify tasks that they find value in completing, rank their priority, and rank their ability to perform them.

SECONDARY OUTCOMES:
Motor evoked potential status (MEPs) | Session 2 (Week 1): Baseline Evaluation, Session 19 (Week 7): Post-intervention Evaluation, Session 21 (Week 15): Follow-up Evaluation
  MEP status is a binary TMS stimulation measure for evaluation of the treatment target or, in this study, corticospinal excitability. There will be an attempt to elicit active MEPs in the biceps, ECR, and FDI. The MEP status of each of the 3 muscles will be tested by finding a hot spot using a single pulse TMS. Individual muscles will be labeled as MEP(-) or MEP(+). The criteria for being MEP(+) is any amplitude present in at least 50% (5/10) of the TMS stimuli using stimulation up to 100% maximal stimulator output.
Maximum Voluntary Contraction (MVC) | Session 2 (Week 1): Baseline Evaluation, Session 19 (Week 7): Post-intervention Evaluation, Session 21 (Week 15): Follow-up Evaluation
  Electromyographic (EMG) recordings will be recorded through surface electrodes secured to th skin over the belly of each muscle. In order to obtain MVCs of each affected upper limb muscle, subjects will perform three contractions of elbow flexion, wrist extension, and finger abduction individually. MVCs will be recorded for 3-5s, separated by ~60s of rest.
H-reflex | Session 2 (Week 1): Baseline Evaluation, Session 19 (Week 7): Post-intervention Evaluation, Session 21 (Week 15): Follow-up Evaluation
  The H-reflex is used to assess the reflexive reaction of the flexor carpi radialis muscle after stimulating the sensory nerve (Ia afferent) fibers. Percutaneous electrical stimulation of the median nerve will be delivered (using 1 ms rectangular electrical stimulus, DS7AH, Digitimer Ltd.) through bipolar electrodes (7-mm stainless steel) just proximal to the elbow. Stimulus intensities will be increased in steps of 0.05 mA, starting below H-reflex threshold and increasing up to measure the H-max and M-max at rest (0.25 Hz). The H-max and Mmax will be measured as peak-to-peak amplitude of the non-rectified response in control subjects and both arms of individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolf SL, Winstein CJ, Miller JP, Taub E, Uswatte G, Morris D, Giuliani C, Light KE, Nichols-Larsen D; EXCITE Investigators. Effect of constraint-induced movement therapy on upper extremity function 3 to 9 months after stroke: the EXCITE randomized clinical trial. JAMA. 2006 Nov 1;296(17):2095-104. doi: 10.1001/jama.296.17.2095. PMID 17077374
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Barreca S, Gowland CK, Stratford P, Huijbregts M, Griffiths J, Torresin W, Dunkley M, Miller P, Masters L. Development of the Chedoke Arm and Hand Activity Inventory: theoretical constructs, item generation, and selection. Top Stroke Rehabil. 2004 Fall;11(4):31-42. doi: 10.1310/JU8P-UVK6-68VW-CF3W. PMID 15592988
- [Background] Benavides FD, Jo HJ, Lundell H, Edgerton VR, Gerasimenko Y, Perez MA. Cortical and Subcortical Effects of Transcutaneous Spinal Cord Stimulation in Humans with Tetraplegia. J Neurosci. 2020 Mar 25;40(13):2633-2643. doi: 10.1523/JNEUROSCI.2374-19.2020. Epub 2020 Jan 29. PMID 31996455
- [Background] Stoykov ME, King E, David FJ, Vatinno A, Fogg L, Corcos DM. Bilateral motor priming for post stroke upper extremity hemiparesis: A randomized pilot study. Restor Neurol Neurosci. 2020;38(1):11-22. doi: 10.3233/RNN-190943. PMID 31609714
- See also: Provides information about current treatment options for stroke patients and their efficacy in helping to restore function of the upper limbs. — https://pubmed.ncbi.nlm.nih.gov/17077374/
- See also: This source describes the Fugl-Meyer evaluation method and how this method has been validated for evaluation of the upper limb. — https://pubmed.ncbi.nlm.nih.gov/1135616/
- See also: This source provides information about the CAHAI evaluation method, specifically about the development of the measure and how the included tests were selected. — https://pubmed.ncbi.nlm.nih.gov/15592988/
- See also: This source outlines a procedure to determine the presence of motor-evoked potentials (MEPs) by transcutaneous magnetic stimulation (TMS) in the upper extremity. This information was used to help us design our protocol. — https://pubmed.ncbi.nlm.nih.gov/31996455/
- See also: This source provides further explanation of the procedure for eliciting motor evoked potentials (MEPs) in the upper extremities. — https://pubmed.ncbi.nlm.nih.gov/31609714/